CLINICAL TRIAL: NCT02827448
Title: Urinary Cell Cycle Arrest Biomarkers as Early Predictors of Acute Kidney Injury Following Advanced Cardiac Replacement Therapies
Brief Title: Effectiveness of NephroCheckTM Test to Predict Acute Kidney Injury Following Advanced Cardiac Replacement Therapies
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BRI - 015-179
Record Dates: First submitted 2015-11-24; First posted 2016-07-11 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Acute Kidney Injury; Heart Failure
Keywords: Left Ventricular Assist Device; Heart Transplantation; Perioperative; Acute Kidney Injury; Renal; Kidney; Total Artificial Heart
MeSH Terms: conditions — Acute Kidney Injury; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test how well the NephroCheckTM Test, a noninvasive laboratory test performed on urine, predicts loss of kidney function in patients that have had a heart transplant or a Left Ventricular Assist Device (LVAD) or Total Artificial Heart (TAH) implanted.

DETAILED DESCRIPTION:
Current strategies for AKI detection rely primarily on elevations in serum creatinine in conjunction with diminished urine output. Unfortunately, deviations in these crude parameters of renal function are largely insensitive and late manifestations of AKI, where acute tubular necrosis has likely already transpired and therefore well beyond the phase where preventive measures may be instituted. Early phase biomarkers, insulin-like growth factor-binding protein 7 ("IGFBP7") and tissue inhibitor of metalloproteinases-2 ("TIMP-2") are critical mediators of G1 cell cycle arrest of renal tubular cells during the early phase of cellular injury, providing a potential therapeutic window to prevent permanent damage. To date, no study has evaluated the efficacy of these early phase renal biomarkers for detecting AKI in advanced heart failure patients undergoing cardiac replacement therapies.

Therefore, the aim of this prospective observational study will be to evaluate the effectiveness of the NephroCheckTM to predict AKI in patients undergoing transplant, LVAD implant, or TAH implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive LVAD or heart transplantation

Exclusion Criteria:

* Patients who are unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have had a heart transplant or LVAD implant.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
[TIMP-2]*[IGFBP7] measurement using NephroCheck following LVAD or TAH implantation | 1 year
Occurrence of AKI following LVAD or TAH implantation | 1 year

SECONDARY OUTCOMES:
[TIMP-2]*[IGFBP7] measurement using NephroCheck following cardiac transplantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Joseph, MD, Principal Investigator — Baylor University
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States

REFERENCES:
- [Background] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670
- [Background] Boyle JM, Moualla S, Arrigain S, Worley S, Bakri MH, Starling RC, Heyka R, Thakar CV. Risks and outcomes of acute kidney injury requiring dialysis after cardiac transplantation. Am J Kidney Dis. 2006 Nov;48(5):787-96. doi: 10.1053/j.ajkd.2006.08.002. PMID 17059998
- [Background] Odim J, Wheat J, Laks H, Kobashigawa J, Gjertson D, Osugi A, Mukherjee K, Saleh S. Peri-operative renal function and outcome after orthotopic heart transplantation. J Heart Lung Transplant. 2006 Feb;25(2):162-6. doi: 10.1016/j.healun.2005.07.011. PMID 16446215
- [Background] Topkara VK, Dang NC, Barili F, Cheema FH, Martens TP, George I, Bardakci H, Oz MC, Naka Y. Predictors and outcomes of continuous veno-venous hemodialysis use after implantation of a left ventricular assist device. J Heart Lung Transplant. 2006 Apr;25(4):404-8. doi: 10.1016/j.healun.2005.11.457. Epub 2006 Feb 28. PMID 16563969
- [Background] Borgi J, Tsiouris A, Hodari A, Cogan CM, Paone G, Morgan JA. Significance of postoperative acute renal failure after continuous-flow left ventricular assist device implantation. Ann Thorac Surg. 2013 Jan;95(1):163-9. doi: 10.1016/j.athoracsur.2012.08.076. Epub 2012 Oct 25. PMID 23103012
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Background] Bihorac A, Chawla LS, Shaw AD, Al-Khafaji A, Davison DL, Demuth GE, Fitzgerald R, Gong MN, Graham DD, Gunnerson K, Heung M, Jortani S, Kleerup E, Koyner JL, Krell K, Letourneau J, Lissauer M, Miner J, Nguyen HB, Ortega LM, Self WH, Sellman R, Shi J, Straseski J, Szalados JE, Wilber ST, Walker MG, Wilson J, Wunderink R, Zimmerman J, Kellum JA. Validation of cell-cycle arrest biomarkers for acute kidney injury using clinical adjudication. Am J Respir Crit Care Med. 2014 Apr 15;189(8):932-9. doi: 10.1164/rccm.201401-0077OC. PMID 24559465
- [Background] Meersch M, Schmidt C, Van Aken H, Martens S, Rossaint J, Singbartl K, Gorlich D, Kellum JA, Zarbock A. Urinary TIMP-2 and IGFBP7 as early biomarkers of acute kidney injury and renal recovery following cardiac surgery. PLoS One. 2014 Mar 27;9(3):e93460. doi: 10.1371/journal.pone.0093460. eCollection 2014. PMID 24675717